CLINICAL TRIAL: NCT05341804
Title: Cognitive and Balance Dual Task Training for People With Schizophrenia - Program System Development and Effectiveness Analysis
Brief Title: Cognitive and Balance Dual Task Training for People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Kaohsiung Medical University (Other); Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20210071
Record Dates: First submitted 2022-04-05; First posted 2022-04-22 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia; Cognition; Balance; Dual Task; Mental Illness; Psychiatric Disorder; Fall Prevention
MeSH Terms: conditions — Schizophrenia; Mental Disorders

STUDY DESIGN:
Intervention Model Description: the cognitive and balance dual task training group (COG&BAL), the balance training group (BAL), and the treatment as usual group
Who Masked: Outcomes Assessor
Masking Description: blinded assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the cognitive and balance dual task training group (Experimental): It is performed using the CogBals software, emphasizing the completion of cognitive tasks while performing balance/strength training during the training process.
  Interventions: Behavioral: cognitive and balance dual task training
- the balance training group (Experimental): Balance/strength training without cognitive challenges.
  Interventions: Behavioral: balance training
- the treatment as usual group (No Intervention): Maintain usual rehabilitation activities.

INTERVENTIONS:
Behavioral: cognitive and balance dual task training — a cognitive and balance dual task training program involving the Internet of Thing technique software - Cognitive and Balance training Simultaneously software
  Other Names: Use Cognitive and Balance training Simultaneously software (CogBals)
  Arms: the cognitive and balance dual task training group
Behavioral: balance training — Includes static balance, dynamic balance and strength training
  Arms: the balance training group

SUMMARY:
After developing and pilot testing the training program, including the CogBals software, a 3-arm, single-blinded, randomized controlled trial is used to recruit 84 participants and then randomly allocated to the cognitive and balance dual task training group (COG&BAL), the balance training group (BAL), and the treatment as usual group. The first two training groups (COG&BAL, BAL) receive training for 60 minutes in a group format, 2 times weekly, for 12 weeks. All participants will be assessed at baseline and posttest. The primary outcome is balance function and secondary outcomes are cognitive functions and the muscular endurance of lower extremities.

DETAILED DESCRIPTION:
Background: Individuals with schizophrenia often experience premature aging and accelerated aging, which increases the challenge of care and recovery. Improvement on balance and implementation of prevention from and deceleration of the disability process is of the critical issues in psychiatric rehabilitation. Unfortunately, evidence- based effective programs are limited. Recently, a novel balance training program through cognitive and balance dual task training has shown better outcomes in the elderly and other clinical populations. Yet, the dual task balance training has not been examined for schizophrenia. This dual task balance training with the Internet of Thing techniques is a novel and important program for middle-aged and older individuals with schizophrenia. Further study is needed to develop the training program and to examine the effectiveness.

Purposes: (1) To develop a cognitive and balance dual task training program involving the Internet of Thing technique software - Cognitive and Balance training Simultaneously software (CogBals software) (1st year); (2) to pilot the feasibility of the balance training program for the middle-aged and older individuals with schizophrenia and revise it (1st year); and (3) to examine the effects of the balance training program on balance, cognitive functions, and the muscular endurance of lower extremities (2nd to 3rd year).

Methods: For the effectiveness analysis phase, a 3-arm, single-blinded, randomized controlled trial is used to recruit 84 participants and then randomly allocated to the cognitive and balance dual task training group (COG&BAL), the balance training group (BAL), and the treatment as usual group. The first two training groups (COG&BAL, BAL) receive training for 60 minutes in a group format, 2 times weekly, for 12 weeks. All participants will be assessed at baseline and posttest. The primary outcome is balance function and secondary outcomes are cognitive functions and the muscular endurance of lower extremities.

Contribution: The study uses cognitive and balance dual task training and expect better outcomes on balance improvement. The program can serve as an evidence- based program to prevent and to decelerate the disability process from people with mental illness. The CogBals software developed by researchers and training in a group format is good to promote in the clinical setting with less manpower.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of schizophrenia or schizoaffective disorder for more than 1 year by psychiatrist according to Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5)
2. age 40-75 years old
3. have stable psychiatric symptoms currently (main psychotropic medications have not been adjusted for two months
4. being able to ambulate independently for more than 10 meters, without a walking device
5. not have significant cognitive impairment (Montreal Cognitive Assessment Taiwan Version, MoCA≧20)
6. can follow study protocol and sign the informed consent form

Exclusion Criteria:

1. currently in the psychiatric acute award
2. currently alcohol or drug use disorder
3. Pregnancy, head trauma and other neuromusculoskeletal injuries affect training safety and compliance
4. intellectual disability
5. Unconsciousness or confusion
6. According to the subject's self-report, those with the following medical history, including severe heart failure, myocardial infarction, angina pectoris, chronic obstructive pulmonary disease, poor blood sugar control (i.e., renal dialysis treatment, diabetic neuropathy or retinopathy), no well-controlled hyperemia: systolic blood pressure> 160 mmHg or diastolic blood pressure> 110 mmHg
7. Currently participating in other interventional study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Mini-Balance Evaluation System Test | Change from baseline at 12 weeks
  score from 0-28; higher score is better
Timed up and go test under single and dual tasks | Change from baseline at 12 weeks
  dual tasks include carrying a cup of water and calculation
Single leg stance test under single and dual tasks | Change from baseline at 12 weeks
  dual tasks include carrying a cup of water and calculation
Chinese version of Activities-specific Balance Confidence Scale | Change from baseline at 12 weeks
  score from 0-100; higher score is better
6 meter walk test | Change from baseline at 12 weeks

SECONDARY OUTCOMES:
Symbol Coding | Change from baseline at 12 weeks
  The participant writes as many answers as possible within 90 seconds.
Digit Span | Change from baseline at 12 weeks
  score from 0-33; higher score is better
Spatial Span | Change from baseline at 12 weeks
  score from 0-32; higher score is better
The Stroop Color and Word Test | Change from baseline at 12 weeks
  The participant reads color words or names ink colors from different pages as quickly as possible within 45 seconds.
Color Trials Test | Change from baseline at 12 weeks
  Color Trials 1 and Color Trials 2
30-second sit to stand test | Change from baseline at 12 weeks
  The participant completes as many full stands as possible within 30 seconds.
Bilateral standing heel-rise test | Change from baseline at 12 weeks
  The participant performs the maximum number of plantar flexions possible, until the point of voluntary fatigue, as fast as possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan